CLINICAL TRIAL: NCT04126278
Title: Calcific Tendonitis Treatment: Barbotage vs. Barbotage With Cortisone Injection: A Randomized Controlled Double-Blind Study
Brief Title: Calcific Tendonitis Treatment: Barbotage vs. Barbotage With Cortisone Injection
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment difficulty.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-01299
Record Dates: First submitted 2019-10-11; First posted 2019-10-15 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Calcific Tendinitis
MeSH Terms: interventions — Dexamethasone; Cortisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Barbotage Injection (Experimental): Subjects receiving barbotage with saline injection
  Interventions: Drug: Barbotage
- Barbotage with Cortisone Injection (Active Comparator): Subjects receiving barbotage with cortisone injection
  Interventions: Drug: Barbotage; Drug: Dexamethasone

INTERVENTIONS:
Drug: Barbotage — Administered as per standard of care
Drug: Dexamethasone — 4 mg of dexamethasone
  Other Names: cortisone
  Arms: Barbotage with Cortisone Injection

SUMMARY:
The purpose of this study is to determine the efficacy of barbotage therapy by comparing the clinical and sonographic changes in patients that solely receive barbotage to patients receiving the standard of care, barbotage with cortisone injection.

DETAILED DESCRIPTION:
Calcific tendonitis is a condition caused by calcium deposits building up in a person's muscles or tendons. If calcium builds up in an area, a person may feel pain and discomfort there. The purpose of this study is to determine the efficacy of barbotage therapy (injecting and washing the shoulder joint with saline) by comparing the amount of pain, shoulder function, and X-Rays in patients with calcific tendonitis that receive the standard of care, barbotage with cortisone injection, against barbotage with saline injection. Receiving barbotage without cortisone is therefore considered experimental.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age and younger than 90 years of age
* Diagnosed with calcific tendonitis and ruled out other shoulder-related pathologies
* Failed 1st line therapy (physical therapy and cortisone injection)

  * Intention to receive barbotage with cortisone as standard of care
  * 3 or more months of shoulder pain
  * Finding of one or more calcifications ≥5 mm in size on either sonogram or radiograph, located on the supraspinatus tendon
  * Positive Hawkin's test or Neer's sign for impingement

Exclusion Criteria:

* Legally incompetent or mentally impaired (e.g. minors, Alzheimer's subjects, dementia, etc.)
* Osteoarthritis of the glenohumeral joint of the affected shoulder
* Previous surgery or barbotage to the affected shoulder
* History of prior allergic/hypersensitivity reactions related to the study medication
* Shoulder instability, glenohumeral arthritis, AC pathology, inflammatory arthropathy, fibromyalgia, frozen shoulder or cervical radiculopathy
* Sub-acromial injection with a corticosteroid or treatment by ESWT during the last 3 months before inclusion
* Younger than 18 years of age or older than 90
* Any patient considered a vulnerable subject

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehul Shah, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Upon reasonable request. Requests should be directed to Mehul.Shah@nyulangone.org. To gain access, data requester will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated early; no participants were enrolled in the Barbotage Injection arm.
Period: Overall Study
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Started | 0 | 4
Completed | 0 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Groups:
- Total: Total of all reporting groups
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection | Total
Number analyzed (Participants) | 0 | 4 | 4
Age, Customized [Mean (Standard Deviation); unit: years]
  Age |  | 65 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation. | 65 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 0 | 2 | 2
  Female | 0 | 1 | 1
  Unknown/Not Specified | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 4 | 4
  Unknown or Not Reported |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 4 | 4
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Score at Visit 1
Description: Pain will be assessed by the Visual Analog Scale which describes pain in terms of no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Time Frame: Visit 1 (Day 0)
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Number analyzed (Participants) | 0 | 4
score on a scale |  | 80 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.

2. Primary Outcome: VAS Score at Visit 2
Description: Pain will be assessed by the Visual Analog Scale which describes pain in in terms of no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Time Frame: Visit 2 (Week 6)
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Number analyzed (Participants) | 0 | 4
score on a scale |  | 75 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.

3. Primary Outcome: VAS Score at Visit 3
Description: Pain will be assessed by the Visual Analog Scale which describes pain in terms or sdlk no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Time Frame: Visit 3 (Month 3)
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Number analyzed (Participants) | 0 | 4
score on a scale |  | 50 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.

4. Primary Outcome: VAS Score at Visit 4
Description: Pain will be assessed by the Visual Analog Scale which describes pain in no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).
Time Frame: Visit 4 (Month 6)
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Number analyzed (Participants) | 0 | 4
score on a scale |  | 60 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.

5. Primary Outcome: QuickDASH Score at Visit 1
Description: Individual's ability to complete tasks, absorb forces, and severity of symptoms are measured by a 11-item QuickDash questionnaire using a 5 point Likert scale. The raw score is the sum of responses and is rescaled into a total score ranging from 0-100; lower scores indicate greater abilities.
Time Frame: Visit 1 (Day 0)
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Number analyzed (Participants) | 0 | 4
score on a scale |  | 31 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.

6. Primary Outcome: QuickDASH Score at Visit 4
Description: as for outcome 5
Time Frame: Visit 4 (Month 6)
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Number analyzed (Participants) | 0 | 4
score on a scale |  | 25 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.

7. Primary Outcome: American Shoulder and Elbow Surgeons (ASES) Index Score at Visit 1
Description: 24-item assessment of pain and daily living related to shoulder conditions. Items are rated on various Likert scales. The raw score is the sum of responses and is converted to a total score. Total scores range from 0 to 100; higher scores indicate a better shoulder condition.
Time Frame: Visit 1 (Day 0)
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Number analyzed (Participants) | 0 | 4
score on a scale |  | 25 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.

8. Primary Outcome: ASES Index Score at Visit 4
Description: as for outcome 7
Time Frame: Visit 4 (Month 6)
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Number analyzed (Participants) | 0 | 4
score on a scale |  | 25 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.

9. Primary Outcome: Radiographic Size of Calcium Deposit at Visit 1
Description: Size of calcium deposit will be assessed with Shoulder X-rays.
Time Frame: Visit 1 (Day 0)
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Number analyzed (Participants) | 0 | 4
centimeters (cm) |  | 43 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.

10. Primary Outcome: Radiographic Size of Calcium Deposit at Visit 4
Description: Size of calcium deposit will be assessed with Shoulder X-rays.
Time Frame: Visit 4 (Month 6)
Population: No patients enrolled in the Barbotage Injection arm (see participant flow).
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
Number analyzed (Participants) | 0 | 4
centimeters (cm) |  | 43 (NA) — According to the study team, there was no difference between the data collected, thus there is no standard deviation.

ADVERSE EVENTS:
Time Frame: 6 months
Description: The total number at risk in the Barbotage Injection arm for Serious Adverse Events, All-Cause Mortality, and Other Adverse events is zero because no participants were enrolled into this arm.
Arm/Group | Barbotage Injection | Barbotage With Cortisone Injection
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 0/0 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT04126278/Prot_SAP_000.pdf